CLINICAL TRIAL: NCT01478542
Title: Improvement of Outcome and Reduction of Toxicity in Elderly Patients with CD20+ Aggressive B-Cell Lymphoma by an Optimised Schedule of the Monoclonal Antibody Rituximab, Substitution of Conventional by Liposomal Vincristine, and FDG-PET Based Reduction of Therapy in Combination with Vitamin D Substitution
Brief Title: OPTIMAL>60 / DR. CHOP, Improvement of Therapy of Elderly Patients with CD20+ DLBCL Using Rituximab Optimized and Liposomal Vincristine
Acronym: OPTIMAL>60
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other); Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL 2009-1
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: CD20+ Aggressive B-Cell Lymphoma
Keywords: DLBCL; Liposomal Vincristine (Marqibo); Optimised Rituximab; Toxicity; Elderly Patients; FDG-PET; Bulky Disease; Radiation; age >60 years; First line Therapy; Vitamin D
MeSH Terms: interventions — Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (6):
- Favourable Prognosis F-A - Recruitment completed (Active Comparator): Induction therapy with 4 cycles of R-CHOP-14 (Rituximab 375 mg/sqm, Cyclophosphamide 750 mg/sqm, Doxorubicin 50 mg/sqm, conventional Vincristine 1,4 mg/sqm [max. 2mg absolute], Predniso[lo]ne 100mg/d d1-5) and then definitive (post-induction) restaging with FDG-PET. If FDG-PET positive 2 additional cycles of R-CHOP-14 + 2xR plus additional involved-site radiotherapy, if FDG-PET negative only 4xR without radiotherapy.
  Interventions: Drug: Conventional Vincristine
- Favourable F-B - Arm Closed (Experimental): Induction therapy with 4 cycles of R-CHLIP-14 (Rituximab 375 mg/sqm, Cyclophosphamide 750 mg/sqm, Doxorubicin 50 mg/sqm, liposomal Vincristine 1,4 mg/sqm (max. 2mg absolute), Predniso[lo]ne 100mg/d d1-5) and then definitive (post-induction) restaging with FDG-PET. If FDG-PET positive 2 additional cycles of R-CHLIP-14 + 2xR plus additional involved-site radiotherapy, if FDG-PET negative only 4xR without radiotherapy.
  Interventions: Drug: Liposomal Vincristine
- Less Favourable LF-A - Recruitment completed (Active Comparator): Induction therapy with 6 cycles of R-CHOP-14 (Rituximab 375 mg/sqm, Cyclophosphamide 750 mg/sqm, Doxorubicin 50 mg/sqm, conventional Vincristine 1,4 mg/sqm [max. 2mg absolute], Predniso[lo]ne 100mg/d d1-5) and then definitive (post-induction) restaging with FDG-PET. If FDG-PET positive 2xR plus additional radiotherapy to the initial bulky region, if FDG-PET negative only 2xR without radiotherapy. After 3xR-CHOP-14 an interim restaging will be performed.
  Interventions: Drug: Conventional Vincristine; Drug: Ricover-scheme rituximab
- Less Favourable LF-B - Recruitment completed (Experimental): Induction therapy with 6 cycles of R-CHLIP-14 (Rituximab 375 mg/sqm, Cyclophosphamide 750 mg/sqm, Doxorubicin 50 mg/sqm, liposomal Vincristine 1,67 mg/sqm [uncapped], , Predniso[lo]ne 100mg/d d1-5) and then definitive (post-induction) restaging with FDG-PET. If FDG-PET positive 2xR plus additional radiotherapy to the initial bulky region, if FDG-PET negative only 2xR without radiotherapy. After 3xR-CHLIP-14 an interim restaging will be performed. Recruitment completed.
  Interventions: Drug: Liposomal Vincristine; Drug: Ricover-scheme rituximab
- Less Favourable LF-C - Recruitment completed (Experimental): Induction therapy with 6 cycles of CHOP-14 (Cyclophosphamide 750 mg/sqm, Doxorubicin 50 mg/sqm, conventional Vincristine 1,4 mg/sqm [max. 2mg absolute], Predniso[lo]ne 100mg/d d1-5) combined with an optimized Rituximab-schedule (375 mg/sqm, d-4, d-1, d1, d4, d14, d28, d42, d56, d91, d126, d175, d238) and then definitive (post-induction) restaging with FDG-PET. If FDG-PET positive additional radiotherapy to the initial bulky region, if FDG-PET negative omission of radiotherapy. After 3x CHOP-14 an interim restaging will be performed. Recruitment completed.
  Interventions: Drug: Conventional Vincristine; Drug: optimised rituximab-schedule
- Less Favourable LF-D - Recruitment completed (Experimental): Induction therapy with 6 cycles of CHLIP-14 (Cyclophosphamide 750 mg/sqm, Doxorubicin 50 mg/sqm, 1,67 mg/sqm [uncapped], , Predniso[lo]ne 100mg/d d1-5) combined with an optimised Rituximab-schedule (375 mg/sqm, d-4, d-1, d1, d4, d14, d28, d42, d56, d91, d126, d175, d238) and then definitive (post-induction) restaging with FDG-PET. If FDG-PET positive additional radiotherapy to the initial bulky region, if FDG-PET negative omission of radiotherapy. After 3x CHLIP-14 an interim restaging will be performed. Recruitment completed.
  Interventions: Drug: Liposomal Vincristine; Drug: optimised rituximab-schedule

INTERVENTIONS:
Drug: Conventional Vincristine
  Arms: Favourable Prognosis F-A - Recruitment completed; Less Favourable LF-A - Recruitment completed; Less Favourable LF-C - Recruitment completed
Drug: Liposomal Vincristine
  Arms: Favourable F-B - Arm Closed; Less Favourable LF-B - Recruitment completed; Less Favourable LF-D - Recruitment completed
Drug: Ricover-scheme rituximab
  Arms: Less Favourable LF-A - Recruitment completed; Less Favourable LF-B - Recruitment completed
Drug: optimised rituximab-schedule
  Arms: Less Favourable LF-C - Recruitment completed; Less Favourable LF-D - Recruitment completed

SUMMARY:
The purpose of this study is to improve the outcome of elderly patients with CD20-Aggressive B-Cell Lymphoma and to reduce the toxicity of standard used Immuno-Chemotherapy by using an optimised schedule of the monoclonal antibody Rituximab, substituting conventional by Liposomal Vincristine and by a PET-guided reduction of therapy in Combination with Vitamin D Substitution.

DETAILED DESCRIPTION:
Primary objective of study:

"OPTIMAL>60 Less Favourable" Patients with less favourable prognosis: To test whether progression-free survival (PFS) can be improved by substituting conventional by liposomal vincristine; To test whether PFS can be improved by 12 optimised applications instead of 8 2-week applications of rituximab.

"OPTIMAL>60 Favourable": Patients with favourable prognosis: Comparison of neurotoxicity of conventional and liposomal vincristine; Determination of PFS for the treatment strategy of reducing treatment in patients with negative FDG-PET after 4 x R-CHOP/CHLIP-14 (PET-4) and comparison with the corresponding patient population in RICOVER-60.

Secondary objectives: "OPTIMAL>60 Favourable" and "OPTIMAL>60 Less Favourable":

Comparison of the prognostic value of a pre-treatment FDG-PET (PET-0) with conventional CT/MRT.

Prospective evaluation on the role of (metabolic) tumor volume to confirm or refuse the hypothesis that optimized rituximab should improve the outcome of patients with a high (metabolic) tumor volume more than that of patients with low MTV and to analyse the substitution of conventional vincristine by liposomal. • Estimation of the vincristine-related neurotoxicity ("OPTIMAL>60 Less Favourable only, since vincristine related neurotoxicity is primary objective of the study in favourable patients") and other toxicities (all patients).

Determination of the therapeutic efficacy of a vitamin D substitution.

Comparison of the FDG-PET-based individualised treatment strategy in OPTIMAL>60 with the fixed (pre-defined) treatment strategy in RICOVER>60.

Investigation of the prognostic value of different FDG-PET derived imaging biomarkers for lymphoma load (SUV, MTV, TLG).

Comparison of the vincristine related neurotoxicity before and after amendment 4.

Comparison of CNS events before and after amendment 4. Comparison of the Cheson, Lugano and RECIL response criteria. Prospective evaluation of the improvement of the prognostic value of ECOG performance status during prephase treatment.

Prospective evaluation of reference pathology biomarkes. Prospective evaluation of circulating tumor DNA (ctDNA), correlation and comparison with PET.

Prospective evaluation of the role of 2 additional cycles of CHOP/CHLIP-14 and involved node radiotherapy in PET-positive patients after 4xR-CHOP/CHLIP-14 in favourable patients.

Evaluation of the role of radiotherapy to PET-positive bulky disease patients after 6xR-CHOP/CHLIP-14 in less favourable patients.

Quality assurance of the performed radiotherapy, including in in-field and outfield relapses.

Investigation of the effect of cross-site ComBat harmonization. Analysis of FDG-PET derived biomarkers in combination with clinical and laboratory variables as distance of lesions and Ann-Arbor stage.

Estimation of the prognostic value of a pre-treatment FDG-PET (PET-0) compared to conventional imaging with CT/MRT.

Prospective evaluation of the prediction of the probability of time-to-progression (TTP) within 2 years by a convolutional neural network trained to analyze maximum intensity projection images from baseline PET.

Analysis regarding molecular subtype, transcriptomics, methylome analysis, spatious analysis of interaction of tumor cells and microenvironment by cyTOF, 3D-morphology (AI-based) or similar techniques, viruses (EBV, HHV6, HHV7), micro-RNA in tumor samples.

Analysis of ctDNA analysis by i) digital droplet PCR, ii) e.g. CAPP or similar methods and iii) methylome analysis as prognostic and predictive marker and comparison with imaging biomarkers.

Analysis special focus on refractory, relapsed courses (including specific patterns of relapse regarding location and time) compared to matched controls and regarding comparison with imaging biomarkers.

Analysis of specific BCR-antigens of aggressive B-NHL as Ars2, SAMD14/neurabin-I in tissue and blood. of initial samples of cases with refractory, relapsing course (including specific patterns of relapse regarding location and time).

Analysis of factors influencing immune effector cells e.g.KIR2DS1 and homozygous HLA-C2, PRF1 A91V or other fHLH variants and prognostic and predictive markers in comparison to RICOVER-60.

Investigation of possible prognostic, or predictive markers of treatment related toxicity as: Neurofilament light chain (NfL) to estimate vincristine-related neurotoxicity, or as clonal hematopoiesis with indeterminate potential (CHIP) and association with cardiovascular events.

Investigation of specific concomitant medication and possible impact on outcome.

Investigation of the efficacy of the modified mandatory infectious prophylaxis OPTIMAL compared to the RICOVER trial with a focus on mandatory chinolon prophylaxis.

Investigation of COVID-19-reated events Impact of interval of diagnosis to time to treatment. Comparison with similar patient populations treated in real-world or prospective clinical trials.

Analysis of EFS and PFS at 24 months (EFS24/PFS24) and its impact on subsequent outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 61-80 years
2. All risk groups (IPI 1-5)
3. Diagnosis of aggressive CD20+ B-NHL, based on an excisional biopsy of a lymph node or on an appropriate sample of a lymph node or of an extranodal involvement. It will be possible to treat the following entities in this study as defined by the new WHO classification of 200870:

   B-NHL:
   * Foll. lymphoma grade IIIb
   * DLBCL, not otherwise specified (NOS)

     * common morphologic variants:

       * centroblastic
       * immunoblastic
       * anaplastic
     * rare morphologic variants
   * DLBCL subtypes/entities:

     * T-cell/histiocyte-rich large B-cell lymphoma
     * primary cutaneous DLBCL, leg type
     * EBV-pos. DLBCL of the elderly
   * DLBCL associated with chronic inflammation
   * primary mediastinal (thymic) LBCL
   * intravascular large B-cell-lymphoma
   * ALK-positive large B-cell-lymphoma
   * plasmoblastic lymphoma
   * primary effusion lymphoma
   * transformed indolent lymphoma secondary or simultaneous high grade B-cell-lymphoma
   * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and Burkitt lymphoma
   * B-cell lymphoma, unclassifiable, with features intermediate between DLCBL and Hodgkin lymphoma
4. Performance status ECOG 0 - 2 after prephase treatment. The performance status of each patient must be assessed before the initiation and after the end of prephase treatment which, as experience has shown, can result in a significant improvement of the patient's performance status. The pre-treatment performance status which can range from ECOG 0 to ECOG 4 must be documented in the Staging CRF (see ISF); the performance status after the prephase treatment must be documented in the respective Prephase Treatment CRF (PT form: see ISF). A definition of the performance status is provided in Appendix 28.10.
5. Written informed consent of the patient
6. Contract of participation signed by the study centre and sponsor

Exclusion Criteria:

1. Already initiated lymphoma therapy (except for the prephase treatment)
2. Serious accompanying disorder or impaired organ function (except when due to lymphoma involvement), in particular:

   * heart: angina pectoris CCS >2, cardiac failure e.g. NYHA >2 and/or EF <50% or FS<25% in nuclear medicine examination/echocardiography
   * lungs: if respiratory problems are suspected the patient is to be excluded if the resultant pulmonary function test shows FeV1<50% or a diffusion capacity <50% of the reference values
   * kidneys: creatinine >2 times the upper reference limit
   * liver: bilirubin >2 times the upper reference limit, aspartate transaminase (AST, SGOT) or alanine transaminase (ALT, SGPT) >3 x institutional upper reference limit
   * uncontrollable diabetes mellitus (prephase treatment with predniso[lo]ne!)
3. Platelets <75 000/mm3, leukocytes <2 500/mm3 (if not due to lymphoma)
4. Known hypersensitivity to the medications to be used
5. Known HIV-positivity
6. Patients with severe impairment of immune defense
7. Patients with constipation with imminent risk of ileus
8. Chronic active hepatitis
9. Poor patient compliance
10. Simultaneous participation in other treatment studies or in another clinical trial within the last 6 months
11. Prior chemo- or radiotherapy, long-term use of corticosteroids or anti-neoplastic drugs for previous disorder
12. Other concomitant tumour disease and/or tumour disease in the past 5 years (except for localised skin tumors other than melanoma and carcinomas in situ of any other origin)
13. CNS involvement of lymphoma (intracerebral, meningeal, intraspinal intradural) or primary CNS lymphoma
14. Persistent neuropathy grade ≥2 (NCI CTC-AE v4.03) (unless due to lymphoma involvement)
15. History of persistent active neurologic disorders grade >2 including demyelinating form of Charcot-Marie-Tooth syndrome, acquired demyelinating disorders, or other demyelinating condition
16. Pregnancy or breast-feeding women
17. Active serious infections not controlled by oral and/or intravenous antibiotics or anti-fungal medication
18. Any medical condition which in the opinion of the investigator places the subject at an unacceptably high risk for toxicities.
19. MALT lymphoma
20. Non-conformity to eligibility criteria
21. Persons not able to understand the impact, nature, risks and consequences of the trial (including language barrier)
22. Persons not agreeing to the transmission of their pseudonymous data
23. Persons depending on sponsor or investigator
24. Persons from highly protected groups. Pts. with CNS lymphoma should not be included in this study.

Ages: 61 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2011-11; Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 9 years
  "OPTIMAL>60 Less Favourable": To test the effects of substitution of conventional by liposomal vincristine and of a 2-week applications of 8x rituximab by an optimised application of 12 x rituximab stratified log rank tests will be performed for each question (stratified for IPI-factors). Proportional hazard models will be used to investigate treatment interaction and to obtain estimates for the single treatment effects (HR) adjusting for the IPI-factors.
  "OPTIMAL>60 Favourable" Grade of neurotoxicity will be estimated and indicated with a 95% confidence interval (CI) separated to each type of vincristine. To investigate the 3-year PFS with 95% CI the Kaplan-Meier estimator will be used.

SECONDARY OUTCOMES:
for efficacy: CR-rate, PR-rate, rate of primary progressions, relapse rate, EFS and OS; rate and CTC grades of PNP. Prognostic value of the FDG-PET derived imaging biomarkers for lymphoma load: SUV, MTV, TLG. | 9 years
  Secondary endpoints: To analyze how (i. e. in which direction) and how often a pre-treatment FDG-PET-based assignment (PET-0) would have affected the assignment of a patient to a different stage, IPI risk group or treatment, respectively. The different FDG-PET derived imaging biomarkers for lymphoma load (SUV, MTV, TLG) will be analyzed for their relationship with CR-rate, PR-rate, rate of primary progressions, relapse rate, EFS, PFS and OS.
  To compare the efficacy and side effects of the (post-induction therapy FDG-PET-based) individualised treatment strategy in OPTIMAL>60 with the fixed (pre-defined) treatment strategy in RICOVER-60.
  Rates and grades of polyneuropathy will be determined according to CTC-v4.03. Comparison of the patients without vitamin-D-substitution with patients receiving a vitamin-D-substitution.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Thurner, Professor, Principal Investigator — Saarland University, Saarland University Hospital
Locations (127):
- Germany (127):
  - Saarland University Hospital, Homburg, Saarland
  - Evangelisches Krankenhaus Paul Gerhardt Stift, Klinik für Innere Medizin II, Wittenberg, Saxony-Anhalt
  - Klinik für Hämatologie und Onkologie, Aachen
  - Innklinikum Altötting, Altötting
  - Klinikum St. Marien Amberg, MVZ, Amberg
  - Klinikum Augsburg, Medizinische Klinik II, Augsburg
  - Praxis Dres. med. Brudler, Heinrich, Bangerter, Augsburg
  - Gemeinschaftspraxis Dres. Reichert, Janssen, Aurich
  - Helios Klinikum Bad Saarow, Klinik für Innere Medizin III, Bad Saarow
  - Sozialstiftung Bamberg, Med. Klinik V, Bamberg
  - Klinikum Bayreuth, Medizinische Klinik IV, Bayreuth
  - Charité- Universitätsmedizin Berlin, Campus Benjamin Franklin, Med. Klinik III, Berlin
  - Knappschaftskrankenhaus Bochum, Bochum
  - Johanniter Krankenhaus Bonn, Abteilung für Innere Medizin I, Bonn
  - Universitätsklinikum Bonn, Med. Klinik III, Bonn
  - Städt. Klinikum Brandenburg, Med. Klinik II, Brandenburg
  - Evangelisches Diakonie-Krankenhaus Bremen, Bremen
  - Praxis Dr. Obst, Burgwedel
  - Praxis Dr. Marquard, Celle
  - Klinikum Chemnitz, Innere Medizin III, Chemnitz
  - Klinikum Coburg, V. Med. Klinik, Coburg
  - Schwerpunktpraxis Dres. Glados/Retzlaff/Zühlsdorf/Deuticke, Coesfeld
  - Gemeinschaftspraxis Dres. Schmitz, Steinmetz, Severin, Cologne
  - Klinikum der Universität zu Köln, Klinik I für Innere Medizin, Cologne
  - Krankenhaus Holweide, Cologne
  - St. Johannes Hospital Dortmund, Med. Klinik II, Dortmund
  - BAG Freiberg-Richter, Jacobasch, Wolf, Illmer, Dresden
  - Gemeinschaftspraxis Dres. Mohm, Prange-Krex, Dresden
  - Universitätsklinikum Erlangen, Med. Klinik 5, Erlangen
  - St.-Antonius-Hospital Eschweiler, Hämatologie und Onkologie, Eschweiler
  - Klinikum Esslingen, Klinik für Gastroenterologie, Onkologie und Innere Medizin, Esslingen am Neckar
  - Klinikum der J.W. Goethe-Universität Frankfurt, Hämatologie/Onkologie, Frankfurt
  - Krankenhaus Nordwest Frankfurt, II. Med. Klinik, Frankfurt
  - Klinikum Frankfurt (Oder), Abteilung f. Innere Medizin, Frankfurt (Oder)
  - Praxis Dr. med. Reiber, Freiburg im Breisgau
  - Universitätsklinikum Freiburg, Innere Medizin I, Freiburg im Breisgau
  - Klinikum Fulda, Med. Klinik III, Fulda
  - St. Josef-Hospital Gelsenkirchen, Onkologie und Hämatologie, Gelsenkirchen
  - Praxis Dr. med. Schliesser, Giessen
  - Wilhelm-Anton-Hospital Goch, Innere Medizin, Goch
  - Onkologische Kooperation Harz, Onkologische Schwerpunktpraxis, Goslar
  - Universitätsmedizin Göttingen, Hämatologie und Onkologie, Göttingen
  - Universitätsmedizin Greifswald, Medizinische Universitätsklinik C, Hämatologie und Onkologie, Greifswald
  - Kreiskrankenhaus Gummersbach, Gummersbach
  - Klinikum Gütersloh, Gütersloh
  - Kath. Krankenhaus Hagen, St.-Marien-Hospital, Hagen
  - Gemeinschaftspraxis Rohrberg, Hurtz, Schmidt, Frank-Gleich, Halle
  - Asklepios Klinik St. Georg, Hämatologie/Onkologie, Hamburg
  - Hämatolog.-onkolog. Praxis Dres. Müller-Hagen, Bertram, Albertinen-Krankenhaus, Hamburg
  - Hämatologisch-onkologische Praxis Altona (HOPA), Hamburg
  - Universitätsklinikum Hamburg-Eppendorf (UKE), II. Med. Klinik und Poliklinik, Onkologie und Hämatologie, Hamburg
  - Klinikum Hannover-Siloah, Klinik für Hämatologie, Hanover
  - Medizinische Hochschule Hannover (MHH), Zentrum für Innere Medizin, Klinik für Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation, Hanover
  - Praxis MediProjekt, Hanover
  - Universitätsklinikum Heidelberg, Innere Medizin V, Heidelberg
  - Klinikum Kreis Herford, Med. Klinik II, Herford
  - Onkologische Schwerpunktpraxis Dres. Freier, Sievers, Hildesheim
  - St. Bernward Krankenhaus Hildesheim, Med. Klinik II, Hildesheim
  - KMT Klinik Idar-Oberstein, Idar-Oberstein
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Jena
  - Westpfalz-Klinikum, Klinik für Innere Medizin I, Kaiserslautern
  - Praxis Dres Hansen, Reeb, Kaiserslautern
  - St. Vincentius Kliniken Karlsruhe, Med. Klinik Abt. 2, Karlsruhe
  - Städtisches Klinikum Karlsruhe, II. Med. Klinik, Hämatologie/Onkologie/Infektionskrankheiten, Karlsruhe
  - GMP Dres Siehl, Söling, Kassel
  - Rotes Kreuz Krankenhaus Kassel, Klinik für Interdisziplinäre Onkologie, Kassel
  - Klinikum Kempten-Oberallgäu, Hämatologie, Onkologie und Palliativmedizin, Kempten
  - Gemeinschaftsklinikum Mittelrhein, Ev. Stift St. Martin, Innere Medizin, Koblenz
  - Gemeinschaftspraxis Dres. Neise, Lollert, Krefeld
  - Praxis Dr. Strauch, Kronach
  - Klinikum Landshut, Med. Klinik I, Landshut
  - Caritas Krankenhaus Lebach, Lebach
  - Onkologische Schwerpunktpraxis, Leer
  - Klinikum St. Georg Leipzig, Abteilung für internistische Onkologie/Hämatologie, Leipzig
  - Klinikum Lippe-Lemgo, Med. Klinik II, Lemgo
  - Onkologische Schwerpunktpraxis Lörrach, Loerrach
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Klinikum Magdeburg, Hämatologie/Onkologie, Magdeburg
  - Universitätsmedizin Mainz, III. Med. Klinik und Poliklinik, Mainz
  - Mannheimer Onkologie Praxis, Dres. Brust, Plöger, Schuster, Hensel, Mannheim
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Johannes Wesling Klinikum, Klinik für Hämatologie, Onkologie und Palliativmedizin, Minden
  - Kliniken Maria-Hilf Mönchengladbach, Innere Medizin I, Mönchengladbach
  - Stauferklinikum Schwäbisch Gmünd, Zentrum für Innere Medizin, Mutlangen
  - GMP Dres Schröder/Sieg, Mülheim
  - Klinikum Großhadern, Med. Klinik 3, München
  - Klinikum rechts der Isar der Technischen Universität München, III. Med.Klinik, München
  - Städtisches Klinikum München Harlaching, München
  - Praxis Dres. Schmidt, Fromm, Wiesmeier, Seufert, Klapthor, Zingerle, München Pasing
  - Universitätsklinikum Münster, Med. Klinik A, Münster
  - Onkologische Praxis Dr. Ladda, Neumarkt
  - Lukaskrankenhaus Neuss, Med. Klinik II, Neuss
  - Kreiskliniken Esslingen, Klinikum Kirchheim-Nürtingen, Hämatologie, Internist. Onkologie und Palliativmedizin, Nürtingen
  - Gemeinschaftspraxis Dres. Balló, Böck, Offenbach
  - Ortenau Klinikum Offenburg-Gegenbach, Medizinische Klinik II, Offenburg
  - Klinikum Oldenburg, Hämatologie/Onkologie, Oldenburg
  - Onkologische Schwerpunktpraxis Dr. Hübner, Oldenburg
  - Pius Hospital Oldenburg, Klinik für Strahlentherapie und Internistische Onkologie, Oldenburg
  - Onkologische Schwerpunktpraxis im MVZ 2 GmbH, Dr. H. Eimermacher, Olpe
  - Klinikum Osnabrück, Med. Klinik III, Osnabrück
  - Paracelsus Krankenhaus Ruit, Kreiskliniken Esslingen gGmbH, Zentrum für Allgemeine Innere Medizin, Ostfildern
  - Brüderkrankenhaus St. Josef Paderborn, Klinik für Hämatologie und Onkologie, Paderborn
  - Gemeinschaftspraxis Dres. Baake, Leonhardt, Moegling, am Regio Klinikum Pinneberg, Pinneberg
  - Klinikum Ernst von Bergmann, Klinik für Hämatologie, Onkologie und Palliativmedizin, Potsdam
  - Gemeinschaftspraxis Dres. Decker, Nonnenbroich, Herbrik-Zipp, Ravensburg
  - Prosper-Hospital Recklinghausen, Med. Klinik I, Recklinghausen
  - Krankenhaus Barmherzige Brüder Regensburg, Klinik für Onkologie und Hämatologie, Regensburg
  - Klinikum am Steinenberg, Kreiskliniken Reutlingen GmbH, Reutlingen
  - Elblandklinikum Riesa, Klinik für Innere Medizin II, Riesa
  - Klinikum Südstadt Rostock, Innere Medizin, Rostock
  - Universitätsklinikum Rostock, Abteilung Hämatologie/Onkologie, Klinik u. Poliklinik für Innere Medizin, Rostock
  - GMP Dres Jacobs, Daus, Schmits, Saarbrücken
  - ZAHO-Siegburg, Zentrum für ambulante Hämatologie und Onkologie Siegburg, Siegburg
  - Diakonie-Klinikum Stuttgart, Med. Klinik II, Stuttgart
  - Klinikum Traunstein, Hämatologie/Onkologie, Traunstein
  - Klinikum Mutterhaus der Borromäerinnen, Med. Abteilung I, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, I. Med. Abteilung, Trier
  - Universitätsklinikum Tübingen, Medizinische Klinik und Poliklinik, Onkologie, Hämatologie, Immunologie und Rheumatologie, Tübingen
  - Universitätsklinikum Ulm, Innere Medizin III, Ulm
  - Katharinen Hospital Unna, Unna
  - Schwarzwald-Baar-Klinikum - Innere Medizin II, Villingen-Schwenningen
  - Praxis Onkologie Schwarzwald - Alb, Villingen-Schwenningen
  - Med. Versorgungszentrum Weiden, Abteilung für Onkologie, Weiden
  - Praxis Dres med. Perker, Sandherr, Weilheim
  - HSK Wiesbaden, Innere Medizin III, Wiesbaden
  - Helios Klinkum Wuppertal, Med. Klinik I, Wuppertal
  - Hämatologisch-Onkologische Praxis Würselen, Würselen

REFERENCES:
- [Background] Pfreundschuh, M., Christofyllakis, K., Altmann, B., Ziepert, M., Haenel, M., Viardot, A., Neubauer, A., Held, G., Truemper, L., Dreyling, M., Kanz, L., Hallek, M., Schmitz, N., Heintges, T., Kölbel, C., Buecker, A., Ruebe, C., Hellwig, D., Berdel, C., Poeschel, V., and Murawski, N. (2017) Radiotherapy to bulky disease PET-negative after immunochemotherapy in elderly DLBCL patients: Results of a planned interim analysis of the first 187 patients with bulky disease treated in the OPTIMAL>60 study of the DSHNHL. Hematological Oncology, 35( S2): 129- 130. doi: 10.1002/hon.2437_119.
- [Derived] Kaddu-Mulindwa D, Altmann B, Held G, Angel S, Stilgenbauer S, Thurner L, Bewarder M, Schwier M, Pfreundschuh M, Loffler M, Menhart K, Grosse J, Ziepert M, Herrmann K, Duhrsen U, Huttmann A, Barbato F, Poeschel V, Hellwig D. FDG PET/CT to detect bone marrow involvement in the initial staging of patients with aggressive non-Hodgkin lymphoma: results from the prospective, multicenter PETAL and OPTIMAL>60 trials. Eur J Nucl Med Mol Imaging. 2021 Oct;48(11):3550-3559. doi: 10.1007/s00259-021-05348-6. Epub 2021 Apr 29. PMID 33928400